CLINICAL TRIAL: NCT05557435
Title: The Effect of Breast Milk Odor on Pain Response and Salivary Cortisol Level Duration Heel Stick Procedure in Preterm Infants: A Randomized Controlled Trial
Brief Title: The Effect of Breast Milk Odor on Pain Response and Salivary Cortisol Level in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: N202204023
Record Dates: First submitted 2022-09-20; First posted 2022-09-28 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-09

CONDITIONS: Premature Infant; Pain; Breast Milk Odor
Keywords: Breast Milk Odor, Pain, salivary cortisol, Preterm Infants, Randomized Controlled Trial
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast milk odor (Experimental): Participants received breast milk odor before and during heel stick.
  Interventions: Other: breast milk odor
- Placebo (Placebo Comparator): Participants received placebo before and during heel stick.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: breast milk odor — The intervention of the experimental group was to stimulate the odor of breast milk. The researchers informed the mothers of premature infants in advance on the day before the experiment, and collected the breast milk samples in the morning before eating on the day of the experiment (excluding the influence of the odor of breast milk by diet). The researchers took a clean cotton ball so that the breast milk was completely absorbed by the cotton ball, and placed the cotton ball that absorbed breast milk at a distance of 5cm next to the mouth and nose of the premature infant, so that the premature infant could receive the smell of breast milk.
  The intervention of the control group was to stimulate the smell of distilled water.
  Arms: Breast milk odor
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aims of this randomized controlled trial are investigate the effects of breast milk odor on pain response and saliva cortisol level duration heel stick blood sampling in preterm infants. Partipants will randomly assigned into the experimental group (breast milk odor) or control group (distilled water odor). The Premature Infant Pain Profile-Revised (PIPP-R) and Salimetrics® Cortisol Enzyme Immunoassay Kit are used to measuring the pain response and saliva cortisol level.

DETAILED DESCRIPTION:
Preterm infants need to undergo more invasive medical interventions than full-term healthy newborns to maintain their lives. Physiological functions changes brought about by pain and stress stimulations may complicate nerve development in preterm infants. Therefore, providing positive sensory supportive interventions to reduce pain and stress is imperative for preterm infants. Studies have confirmed that the use of painkillers, breastfeeding, swaddling, kangaroo care, giving glucose or sucrose can help reduce pain. The sense of smell matures at 28 weeks of gestation age, and newborns can recognize the mother's smell after birth (Nishitani et al., 2009).

In recent years, several randomized studies have explored the effects of smell on reducing pain and stress in preterm infants, but the results are still inconclusive due to the lack of randomization blinding and a variety of smell interventions. It is desirable to plan a high-quality study. Although premature infants need to be separated from their mothers in nurseries due to medical needs, breast milk is still the best source of nutrition. The aims of this study are to investigate the effect of breast milk odor on pain response and saliva cortisol level duration heel stick blood sampling in preterm infants with gestation age at 30 to 37 weeks. A Randomized Controlled Trial will be designed. Preterm infants, who will receive heel sticks, are randomly assigned into the experimental group (breast milk odor) or control group (distilled water odor). The Premature Infant Pain Profile-Revised (PIPP-R) and Salimetrics® Cortisol Enzyme Immunoassay Kit are used to measuring the pain response and saliva cortisol level. Data will be analyzed by SPSS 22.0 (SPSS Inc., Chicago, IL, USA) using descriptive statistics, independent t-test, ANOVA, Generalized Estimating Equation linear multiple regression analysis… etc.

ELIGIBILITY:
Inclusion Criteria:

1. Premature babies whose gestational age is between 30 weeks to 36 weeks and six days, with a birth weight > 1000 grams.
2. Apgar Score > 6 at 5 minutes of birth.
3. Within 10 days of birth, the vital signs are stable.
4. Those who have medical needs, such as blood monitoring of neonatal serum bilirubin, blood sugar, electrolyte, or neonatal screening, etc., need heel puncture blood sampling.

Exclusion Criteria:

1. Those who have been diagnosed by a physician with severe congenital malformations, chromosomal abnormalities, respiratory distress, epilepsy, necrotizing enterocolitis, intracranial hemorrhage, periventricular leukomalacia, sepsis, meningitis, or hyperbilirubinemia.
2. Those who have bronchopulmonary dysplasia or other chronic lung diseases that require the use of ventilator or non-invasive positive pressure respiratory support.
3. Have used analgesics or anesthetics within 48 hours before giving the intervention of the study, or are participating in other studies that provide intervention for pain reduction.

Ages: 0 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain on PIPP-R(Premature Infant Pain Profile - Revised, PIPP-R) in experimental group and control group from baseline and the time during heel stick. | before heel stick [baseline] and during heel stick [5th minute].
  PIPP-R is suitable for newborns from GA 25 to 41 weeks. The evaluation items include: two physiological indicators (heartbeat, blood oxygen), three behavioral indicators (frowning, closed eyes, facial expressions such as nasolabial folds), and two corrections factors (gestational weeks and behavioral status). Each item is scored on a scale of 0 to 3 on four scales. The full score varies according to the gestational week: 21 points up to 28 weeks, 20 points for 28 to 31+6 weeks, 19 points for 32 to 35+6 weeks, and 18 points for over 36 weeks. A total PIPP-R score of 6 or less indicates little or no pain, a score of 6 to 12 indicates mild to moderate pain, and a score greater than 12 indicates moderate to severe pain.
Change in salivary cortisol in experimental group and control group from baseline to the time after heel stick. | before heel stick [baseline] and 25 minutes after heel stick [30th minute, reflecting pain and stress conditions at the moment of heel stick])
  Salimetrics® Cortisol Enzyme Immunoassay Kit Analytical sensitivity .Salivary cortisol samples in neonatal detection range: not detected to 3.41μg/dL.